CLINICAL TRIAL: NCT03142607
Title: Comparative Evaluation of Chlorhexidine, Metronidazole and Combination Gels on Gingivitis: A Randomized Clinical Trial
Brief Title: Comparative Evaluation of Chlorhexidine, Metronidazole and Combination Gels on Gingivitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Sheikh Bilal Badar, Resident Investigator, Aga Khan University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4577-Sur-ERC-16
Record Dates: First submitted 2017-04-28; First posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — chlorhexidine gluconate

STUDY DESIGN:
Intervention Model Description: Group A has Metronidazole gel Group B has Chlorhexidene gel Group C has combination of metronidazole and chlorhexidene gel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will be assigned to one of the three study groups using a computer generated randomization list. The recruitment of the patients will be performed by one investigator. All the measurements at the baseline and follow ups will be performed by the second investigator. Patient, the care provider, the investigator who is taking the measurement and the statistician will be blinded about the intervention groups. This will be ensured by giving codes to the intervention groups only known to the principal investigator who is not involved in the measurement and interaction with the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): subjects will be instructed to apply a standard 0.2 % Chlorhexidine gel (clinica gel) on the marginal gingiva for the next 14 days, twice a day for 30 minutes, after morning and evening tooth brushing
  Interventions: Drug: Chlorhexidine Gluconate
- Group B (Active Comparator): Subjects will be instructed to apply 0.8 % Metronidazole gel (anaerobic gel) twice daily for 30 minutes after morning and evening tooth brushing for two weeks
  Interventions: Drug: Metronidazole gel
- Group C (Active Comparator): subjects will be instructed to apply 0.2 % Chlorhexidine gel (clinica gel) on the marginal gingiva after morning tooth brushing for 30 minutes and 0.8 % metronidazole gel (anaerobic gel) after evening tooth brushing for 30 minutes for two weeks. Subjects in these groups will receive the detailed and precise instruction and demonstrations on the diurnal alternate application of the two gels
  Interventions: Drug: Metronidazole gel; Drug: Chlorhexidine Gluconate

INTERVENTIONS:
Drug: Metronidazole gel — 1% Metronidazole gel
  Other Names: Revomet gel
  Arms: Group B; Group C
Drug: Chlorhexidine Gluconate — 0.2% Chlorhexidene gluconate gel
  Other Names: Clinica gel
  Arms: Group A; Group C

SUMMARY:
Patient presenting to the dental clinic with gingivitis and fulfilling the inclusion criteria will be included in the study after taking informed consent. Participants will be divided into three groups. Each group will be instructed to apply metronidazole gel, chlorhexidine gel or combination of metronidazole and chlorhexidine gel on the marginal gingiva. Measurement for the gingival index will be taken at baseline, at 2 weeks and at 4 weeks interval

DETAILED DESCRIPTION:
Training of the examiner:

Participating investigators(Resident and supervisor) will be trained and calibrated on the development of the trial, case selection, measurement techniques, sample collection, data compilation sheets and their precise role in the study. In order to evaluate the intra-examiner reliability, five subjects not involved in the study will be evaluated twice by each investigator for the measurements at the interval of one week.

Methodology:

On the first visit after clinical examination, the specially designed baseline study proforma will be filled-in. The bleeding sites, probing depth and the gingival index score will be calculated.

Group A subjects will be instructed to apply a standard 0.2 % Chlorhexidine gel (clinica gel) on the marginal gingiva for the next 14 days, twice a day for 30 minutes, after morning and evening tooth brushing.

Group B subjects will be instructed to apply 0.8 % Metronidazole gel (anaerobic gel) twice daily for 30 minutes after morning and evening tooth brushing for two weeks.

Group C subjects will be instructed to apply 0.2 % Chlorhexidine gel (clinica gel) on the marginal gingiva after morning tooth brushing for 30 minutes and 0.8 % metronidazole gel (anaerobic gel) after evening tooth brushing for 30 minutes for two weeks. Subjects in these groups will receive the detailed and precise instruction and demonstrations on the diurnal alternate application of the two gels.

The application of the topical gels will be halted after 2 weeks and second clinical examination will be carried out for bleeding sites, probing depth and the gingival index score. Scaling & polishing of teeth in all three groups and oral hygiene instructions will be reinforced. Subjects will be recalled at 4 week for evaluation of gingival and oral hygiene indices. The reading will be recorded in the study proforma.

Randomization, blinding and treatment allocation:

Subjects will be assigned to one of the three study groups using a computer generated randomization list. The recruitment of the patients will be performed by one investigator. All the measurements at the baseline and follow ups will be performed by the second investigator. Patient, the operator (until the gel will be handed over by the dental assistant), the investigator who is taking the measurement and the statistician will be blinded about the intervention groups. This will be ensured by giving codes to the intervention groups only known to the principal investigator who is not involved in the measurement and interaction with the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients having 20 or more healthy teeth
* Systematically healthy patient with no co-morbid
* Subjects with clinically confirmed gingivitis having positive bleeding gums on probing in every sextant
* Subjects having teeth without any clinical attachment loss

Exclusion criteria:

* Subjects with clinical attachment loss of greater than 2 mm on two sites
* Pregnant or lactating females
* Subjects with removal or fixed dental prosthesis
* History of surgical or nonsurgical periodontal therapy in the last 6 months
* Use of antibiotic in the last 30 days
* Habit of smoking or use of smokeless tobacco
* Allergic to Metronidazole or Chlorhexidine
* Presence of any craniofacial syndrome patients
* Patients on medications that have effects on gingival conditions (such as Nifedipine, Cyclosporine and Phenytoin etc.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-02-03 (Actual); Primary Completion 2018-01-02 (Estimated); Study Completion 2018-02-02 (Estimated)

PRIMARY OUTCOMES:
Change in Gingival Index | Two weeks and four weeks
  On each appointment, gingival index values will be evaluated and change in the gingival index will be noted.

SECONDARY OUTCOMES:
Change in Oral Hygiene Index | Two weeks and four weeks
Change in Bleeding index | Two weeks and four weeks
Change in Probing depth | Two weeks and four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robia Ghafoor, BDS, FCPS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No